CLINICAL TRIAL: NCT00468117
Title: Islet Transplantation in Type 1 Diabetic Kidney Allograft Recipients: Efficacy of Islet After Kidney Transplantation (CIT-06)
Brief Title: Efficacy of Islet After Kidney Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CIT-06
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Hypoglycemia; Kidney Transplant; Insulin independence; Islet Transplantation; Intensive Insulin Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Islets of Langerhans Transplantation; Antilymphocyte Serum; Daclizumab; Basiliximab; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Islet transplantation (Experimental): Up to three separate islet transplants will occur and a regimen of immunosuppressive medications consisting of antithymocyte globulin (ATG) and etanercept throughout study.
  Interventions: Procedure: Islet transplantation; Biological: Antithymocyte Globulin; Biological: Daclizumab or Basiliximab; Biological: Etanercept; Biological: Allogenic human purified pancreatic islets

INTERVENTIONS:
Procedure: Islet transplantation
Biological: Antithymocyte Globulin — Participants will begin receiving ATG 2 days prior to the initial islet transplant and will continue to receive ATG until Day 2 post-transplant.
  Other Names: ATG
Biological: Daclizumab or Basiliximab — Daclizumab or Basiliximab will be used for subsequent transplants.
Biological: Etanercept — Etanercept will be given on the day of transplant and on Days 3, 7, and 10 post-transplant.
Biological: Allogenic human purified pancreatic islets — 200 ml suspension of allogenic human purified islets

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the insulin-producing pancreatic beta cells are destroyed, resulting in poor blood sugar control. The purpose of this study is to assess the benefit of islet transplantation in type 1 diabetic (T1D) kidney transplant recipients.

DETAILED DESCRIPTION:
Type 1 diabetes is commonly treated with the administration of insulin, either by multiple insulin injections or by a continuous supply of insulin through a wearable pump. Insulin therapy allows long-term survival in individuals with type 1 diabetes; however, it does not guarantee constant normal blood sugar control. Because of this, long-term type 1 diabetic survivors often develop vascular complications, such as diabetic retinopathy, an eye disease that can cause poor vision and blindness, and diabetic nephropathy, a kidney disease that can lead to kidney failure and thus kidney transplant. Some individuals with type 1 diabetes develop hypoglycemia unawareness, a life-threatening condition that is not easily treatable with medication and is characterized by reduced or absent warning signals for hypoglycemia. For such individuals, pancreas or pancreatic islet transplantation are possible treatment options. The purpose of this study is to assess the benefit of islet transplantation in type 1 diabetic kidney transplant recipients.

Participants in this study will be type I diabetics who have received a kidney transplant for ESRD.. If subjects have not received ITT in the 12 months prior to enrollment, they must undergo a period of standardized diabetes care by an experienced diabetologist at the transplant center using the current ADA's standards of medical care in diabetes. Throughout the study, all participants will remain on the immunosuppressive therapy intended for their kidney. Participants will receive up to three separate islet transplants and a regimen of immunosuppressive medications consisting of antithymocyte globulin (ATG) and etanercept. They will begin receiving ATG 2 days prior to transplant and will continue to receive ATG until Day 2 post-transplant. Etanercept will be given on the day of transplant and on Days 3, 7, and 10 post-transplant.

Transplantations will involve an inpatient hospital stay and infusion of islets into a branch of the portal vein. Participants who do not achieve or maintain insulin independence by Day 30 post-transplant will be considered for a second islet transplant. Participants who remain dependent on insulin for longer than 30 days after the second transplant and who show partial graft function will be considered for a third islet transplant. Daclizumab will be used in place of ATG for the second and third transplants, if they are necessary. Participants who do not meet the criteria for a subsequent transplant will enter a reduced follow-up period.

There will be approximately 15 study visits. A physical exam, review of adverse events, and blood collection will occur at most visits. A chest x-ray, abdominal ultrasound, electrocardiogram, quality of life questionnaires, and urine collection will occur at some visits. Participants will also test their own blood glucose levels throughout the study. A 36-month follow-up period will take place after the participant's last transplant, consisting of 8 additional visits.

ELIGIBILITY:
Inclusion Criteria:

* Mentally stable and able to comply with study procedures;
* Clinical history compatible with type 1 diabetes with onset of disease at less than 40 years of age, insulin dependence for at least 5 years at study entry, and a sum of age and insulin dependent diabetes duration of at least 28;
* Absent stimulated C-peptide (defined as less than 0.3 ng/ml) 60 and 90 minutes post-mixed-meal tolerance test;
* Received kidney transplant for ESRD and are taking appropriate calcineurin inhibitor (CNI) based maintenance immunosuppressive therapy;
* Stable renal function as defined as creatinine of no more than one third greater than the average creatinine determination performed in the 3 previous months prior to islet transplantation, until rejection, obstruction or infection is ruled out;
* Intensive diabetes management followed by reduced awareness of hypoglycemia or an HbA1c ≥ 7.5%.

Exclusion Criteria:

* Body mass index (BMI) greater than 30 kg/m2 or weight more than 90 kg;
* Insulin requirement of >1.0 IU/kg/day or <15 U/day;
* Other (non-kidney) organ transplants except prior failed pancreatic graft where the graft failed within the first two weeks due to thrombosis, followed by pancreatectomy and the pancreas transplant occurred more than 6 months prior to enrollment;
* Untreated proliferative diabetic retinopathy;
* Systolic blood pressure higher than 160 mmHg or diastolic blood pressure higher than 100 mmHg;
* Calculated glomerular filtration rate of less than 40 ml/min/1.73meter-squared. More information about this criterion is in the protocol;
* Proteinuria (albumin/creatinine ratio or ACr > 300 mg/g) of new onset since kidney transplantation;
* Either Class I or Class II panel-reactive anti-HLA antibodies > 50%; Participants with either Class I or Class II panel reactive anti-HLA antibodies of 50% or less will be excluded if any of the following are detected:

  1. Positive cross match;
  2. Islet donor-directed anti-HLA antibodies detected my Luminex Single Antigen/specificity bead assay, including weakly reactive antibodies that would not be detected by a flow cross-match; or
  3. Antibodies to the renal donor (i.e. presumed de novo).
* Pregnant, breastfeeding, or unwilling to use effective contraception throughout the study and 4 months after study completion;
* Active infection, including hepatitis B, hepatitis C, HIV, or tuberculosis. More information about this criterion is in the protocol.
* Negative for Epstein-Barr virus (EBV) by (VCA) IgG determination;
* Invasive aspergillus infection, histoplasmosis, and coccidioidomycosis infection one year prior to study enrollment;
* History of malignancy except for completely resected squamous or basal cell carcinoma of the skin;
* Known active alcohol or substance abuse;
* History of Factor V Leiden mutation;
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy after transplantation or individuals with an INR greater than 1.5;
* Severe co-existing cardiac disease, characterized by any one of these conditions:

  1. Recent MI (within past 6 months);
  2. Evidence of ischemia on functional cardiac exam within the last year;
  3. Left ventricular ejection fraction < 30%; or
  4. Valvular disease requiring replacement with prosthetic valve.
* Persistent elevation of liver function tests at the time of study entry. Persistent serum glutamic-oxaloacetic transaminase (SGOT [AST]), serum glutamate pyruvate transaminase (SGPT [ALT],) alkaline phosphatase or total bilirubin, with values > 1.5 times normal upper limits will exclude a subject;
* Active infections (except mild skin and nail fungal infections);
* Acute or chronic pancreatitis;
* Active peptic ulcer disease, symptomatic gallstones, or portal hypertension;
* Treatment with any anti-diabetic medication other than insulin within the past 4 weeks;
* Use of any investigational agents within the past 4 weeks;
* Received live attenuated vaccine(s) within the past 2 months;
* Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial;
* Male participants with elevation of prostate specific antigen (PSA) of more than 4 unless cancer has been excluded;
* Any condition other than T1D as the primary cause of end stage renal disease (ESRD) in the native kidney;
* Positive screen for BK virus by polymerase chain reaction (PCR) determination at time of screening;
* A previous islet transplant;
* A kidney transplant recipient with T1D who has an HbA1c < 7.5% and no history of severe hypoglycemia.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-01; Primary Completion 2015-07 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients w/HbA1c </= to 6.5% and an absence of severe hypoglycemic events or a reduction in HbA1c of at least 1 point and an absence of severe hypoglycemic events | At 1 year after first islet infusion

SECONDARY OUTCOMES:
Reduction in insulin requirements, HbA1c, MAGE, LI, HYPO score, fasting glucose, beta score, serum creatinine, c-peptide levels, MMTT, Clarke Survey, FSIGT, CGMS, number of hypoglycemic events, renal impact, cardiovascular impact, and quality of life | At 1 year after first islet infusion and/or 1 year after final islet infusion

CONTACTS AND LOCATIONS:
Overall Officials: James F. Markmann, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (10):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Emory Universtiy, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Clinical Islet Transplantation Consortium website — http://www.citisletstudy.org